CLINICAL TRIAL: NCT01621321
Title: A Randomized Controlled Trial of Voriconazole in Allergic Bronchopulmonary Aspergillosis
Brief Title: Voriconazole Versus Oral Steroids in Allergic Bronchopulmonary Aspergillosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Cipla Ltd. (Industry)
Responsible Party: Principal Investigator, Ritesh Agarwal, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABPA/003
Record Dates: First submitted 2012-06-12; First posted 2012-06-18 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Prednisolone; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid group (Experimental)
  Interventions: Drug: Prednisolone
- Voriconazole group (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Prednisolone — Prednisolone 0.5 mg/kg/day for 4 weeks; 0.25 mg/kg/day for 4 weeks; 0.125 mg/kg/day for 4 weeks. Then taper by 5 mg every 4 weeks and discontinue. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) 1 puff BD and as needed as per the SMART approach for control of asthma
  Arms: Steroid group
Drug: Voriconazole — Voriconazole 200 mg BD for 4 months. Patients will also receive inhaled formoterol/fluticasone (6/125 mcg) 1 puff BD and as needed as per the SMART approach for control of asthma
  Other Names: Voritek 200 mg twice daily for four months
  Arms: Voriconazole group

SUMMARY:
This is a research project to evaluate the efficacy and safety of two different treatment protocols in Allergic bronchopulmonary Aspergillosis.

DETAILED DESCRIPTION:
Allergic bronchopulmonary aspergillosis (ABPA) is a pulmonary disorder caused by a complex hypersensitivity response to antigens released by the fungus Aspergillus fumigatus. The management of ABPA includes two important aspects - institution of immunosuppressive therapy in the form of glucocorticoids to control the immunologic activity, and close monitoring for detection of relapses. Another possible target is to use antifungal agents to attenuate the fungal burden secondary to the fungal colonization in the airways. Oral corticosteroids are currently the treatment of choice for ABPA associated with bronchial asthma.They not only suppress the immune hyperfunction but are also anti-inflammatory. However, there is no data to guide the dose and duration of glucocorticoids and different regimens of glucocorticoids have been used in literature.Itraconazole, an oral triazole with relatively low toxicity, is active against Aspergillus spp. in vitro and in vivo. The activity of itraconazole against Aspergillus spp. is more than that of ketoconazole. The administration of itraconazole can eliminate Aspergillus in the airways and can theoretically reduce the allergic responses in ABPA. The new triazoles, such as voriconazole, have recently been found effective in the treatment of fungal infections. The investigators hypothesize that voriconazole might also be useful in the treatment of ABPA. The aim of this prospective randomized controlled trial (RCT) is to evaluate the efficacy and safety of voriconazole therapy in patients with ABPA.

ELIGIBILITY:
Inclusion Criteria:

Presence of all the following three criteria:

* Immediate cutaneous hyperreactivity on aspergillus skin test
* Elevated total IgE levels > 1000 IU/mL
* A fumigatus specific IgE levels > 0.35 kUA/L

And, two of the following criteria:

* Presence of serum precipitating antibodies against A fumigatus
* Fixed or transient radiographic pulmonary opacities
* Total eosinophil count > 1000/µL
* Central bronchiectasis on HRCT

Exclusion Criteria:

* Failure to give informed consent
* Intake of glucocorticoids for more than three weeks in the preceding six months
* Enrollment in another trial of ABPA
* Any exposure to azoles in the last six months

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Response rates in the two groups | Six weeks and three months
  IgE levels decline by >=25 percent and there is clinical improvement with partial/total clearance of chest radiographic lesions [if pulmonary opacities have been previously present] after six and three months of treatment
Relapse rates in the two groups | 12, 18, 24 months
  No ABPA exacerbations over the next 3 months after stopping therapy

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 4 months
  Adverse events in the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

REFERENCES:
- [Derived] Agarwal R, Dhooria S, Sehgal IS, Aggarwal AN, Garg M, Saikia B, Chakrabarti A. A randomised trial of voriconazole and prednisolone monotherapy in acute-stage allergic bronchopulmonary aspergillosis complicating asthma. Eur Respir J. 2018 Sep 18;52(3):1801159. doi: 10.1183/13993003.01159-2018. Print 2018 Sep. No abstract available. PMID 30049743